CLINICAL TRIAL: NCT00834015
Title: Outcome of Lumbar Spinal Fusion Patients and Significance of Postoperative Exercise Therapy: Randomized Controlled Trial and Spine Register Study
Brief Title: Spinal Fusion and Rehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jyväskylä Central Hospital (Other)
Collaborators: Tampere University Hospital (Other); Tampere University (Other)
Responsible Party: Principal Investigator, Arja Häkkinen, Professor, Jyväskylä Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Ksshp Dnro 4E/2008; Ksshp Dnro 4E/2008 (Other: K-Sshp)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Spondylolisthesis, Degenerative; Spondylolisthesis, Isthmic
Keywords: spinal fusion; pain; disability; muscle strength; mobility; quality of life; lumbar; isthmic or degenerative spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Other): combined strength and aerobic training
  Interventions: Other: Outcome of lumbar spinal fusion patients and significance of postoperative exercise therapy: A randomized controlled trial

INTERVENTIONS:
Other: Outcome of lumbar spinal fusion patients and significance of postoperative exercise therapy: A randomized controlled trial — combined strength and aerobic training group
  Other Names: Intervention group

SUMMARY:
The aim of the present study is to analyse the significance of postoperative combined strength and aerobic training for outcome of the lumbar fusion patients compared to usual care (patients with isthmic or degenerative spondylolisthesis).

DETAILED DESCRIPTION:
Most of the studies published so far about lumbar fusion surgery have been interested in surgical procedure itself or in comparison of conservative or operative treatment. Less information is available about long-term outcome and exercise programs for operated patients. Therefore the investigators have developed "Spine fusion register", which include data on surgery procedure and outcome (pain, disability, back muscle function, quality of life, working capacity, reoperations and complications etc.) before and after surgery up to 5 years (started in January 1st, 2008). The main purpose of the present study is to analyze the significance of 12-month strength and aerobic training for outcome of the lumbar fusion patients compared to usual care. Patients (N=100) with lumbar fusion because of isthmic or degenerative olisthesis will be will be stratified by catchments area and randomized into combined strength and aerobic training group or into the control group.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* isthmic or degenerative spondylolisthesis

Exclusion Criteria:

* cardiovascular or musculoskeletal diseases, which may exclude their ability to perform strength and endurance training and testing
* metabolic bone disease
* psychosocial instability
* malignant disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
pain | baseline, 1 year (+ 1 year follow-up)
  visual analogue scale (VAS)
disability | baseline, 1 year (+ 1 year follow-up)
quality of life | baseline, 1 year (+ 1 year follow-up)

SECONDARY OUTCOMES:
trunk muscle strength | baseline, 1 year
  isometric strength of flexor and extensor
spine mobility | baseline, 1 year
  flexion tests and lateral bending test
fear of movement | baseline, 1 year postoperatively
  Tampa Scale for Kinesiophobia
physical activity | baseline, 1 year
  International Physical Activity Questionnaire (short form)
depressive symptoms | baseline, 1 year
  DEPS-scale

CONTACTS AND LOCATIONS:
Overall Officials: Arja Häkkinen, Professor, Study Director — Department of Health Sciences, University of Jyväskylä; Marko Neva, Phd, MD, Principal Investigator — Tampere University Hospital; Keijo Häkkinen, professor, Principal Investigator — Department of Biology of Physical Activity, University of Jyväskylä; Joost Dekker, professor, Principal Investigator — Department of Rehabilitation Medicine, VU University Medical Center, Amsterdam, the Netherlands; Kimmo Vihtonen, Phd, MD, Principal Investigator — Department of Surgery, University of Tampere; Outi Ilves, Msc, PT, Principal Investigator — Department of Health Sciences University of Jyvaskyla
Locations (1):
- Jyväskylä Central Hospital, Jyväskylä, Finland

REFERENCES:
- [Derived] Tarnanen S, Neva MH, Dekker J, Hakkinen K, Vihtonen K, Pekkanen L, Hakkinen A. Randomized controlled trial of postoperative exercise rehabilitation program after lumbar spine fusion: study protocol. BMC Musculoskelet Disord. 2012 Jul 20;13:123. doi: 10.1186/1471-2474-13-123. PMID 22817607